CLINICAL TRIAL: NCT03402100
Title: Eye Drops Study for Myopia Control in Schoolchildren
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 103-3476A3
Record Dates: First submitted 2018-01-04; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Myopia, Progressive; Atropine Allergy
Keywords: myopia; schoolchildren; atropine; allergy; eye drops; outdoor; near work
MeSH Terms: conditions — Myopia, Degenerative; Myopia; Hypersensitivity | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.01% atropine (Experimental): children who received 0.01% atropine for myopia
  Interventions: Drug: eye drops
- 0.005% atropine (Experimental): children who received 0.005% atropine for myopia
  Interventions: Drug: eye drops
- 0.25% Ketorolac (Experimental): children who received 0.25% Ketorolac for myopia
  Interventions: Drug: eye drops
- 0.01% atropine plus 0.25% Ketorolac (Experimental): children who received 0.01% atropine plus 0.25% Ketorolac for myopia
  Interventions: Drug: eye drops
- 0.005% atropine plus 0.25% Ketorolac (Experimental): children who received 0.005% atropine plus 0.25% Ketorolac for myopia
  Interventions: Drug: eye drops

INTERVENTIONS:
Drug: eye drops — children who received daily eye drops for myopia

SUMMARY:
The myopia prevalence in schoolchildren is high in Taiwan. The myopia progression is fast in children and often associated high myopia in later life. This prospective and randomized study to investigate the effect of myopia control in myopic children with ultra low concentrations of atropine eye drops and/or low concentrations of anti-allergic and inflammatory eye drops.

DETAILED DESCRIPTION:
Myopia onset earlier in children who would suffer a high degree of myopia in the future adulthood.and higher risk for retinal detachment, macular degeneration, and even blindness. In Taiwan, myopia macular degeneration is the first place of irreversible blind cause in the elderly. The evidence based medicine shows atropine is the most effective treatment for the progression of myopia so far, but the side effects including photophobia and near blurred vision often disturbing patients and resulting poor compliance and high drop-out rate.

Recently, the studies from Taiwan and Singapore showed that low concentrations of atropine (0.05% or 0.01%) can effectively inhibit the myopia progression, reduce the symptoms of photophobia, and to achieve favorable myopia control. Previous study found that myopia and allergic conjunctivitis and inflammation were related. The investigators designed a prospective and randomized study to investigate the effect of myopia control in myopic children with ultra low concentrations of atropine eye drops and/or low concentrations of anti-allergic and inflammatory eye drops. Due to environmental factors such as near work, after school class and outdoor activity are also great associated with myopia, the questionnaires also are collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Myopia diagnosed with the spherical equivalent refraction at least -0.5 diopter (D)
* Must be able to use eye drops

Exclusion Criteria:

* astigmatism -1.50 D or greater
* strabismus
* amblyopia
* cataract
* glaucoma
* any ocular diseases ocular surgery
* history of systemic diseases (ex. asthma, heart disease...)
* contact lenses user
* orthokeratology user

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2014-10-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic spherical refraction change measured by auto-refractometer (Diopter) | 1 year
  Cycloplegic spherical refraction change measured by auto-refractometer (Diopter) is the main indicator of the myopia progression.
Axial length change (mm) measured by non-contact biometry | 1 year
  Axial length change (mm) measured by non-contact biometry is another indicator of the myopia progression.

SECONDARY OUTCOMES:
Intraocular pressure (mmHg) by non-contact tonometer | 1 year
  measures Intraocular pressure (mmHg) by non-contact tonometer
Accommodation (diopter) by accommodometer | 1 year
  Accommodation change (diopter) by accommodometer is another indicator of the myopia progression.
Pupil size (mm) by electronic rule | 1 year
  measures Pupil size (mm) by electronic rule
Anterior chamber depth (mm) measured by non-contact biometry | 1 year
  measures Anterior chamber depth (mm) measured by non-contact biometry
Posterior chamber depth (mm) measured by non-contact biometry | 1 year
  measures Posterior chamber depth (mm) measured by non-contact biometry

OTHER OUTCOMES:
Questionnaire | 1 year
  Record by patients and their parents about how many hours per week of near work (ex. computer/video game,cell phone,reading, piano playing...) and outdoor activities, the compliance of atropine use, discomfort after atropine use (ex. photophobia or blurred vision when near work)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chang Wu, MD, Principal Investigator — No.123,DAPI Rd. Niaosong Dist, Kaohsiung City 83301 Taiwan, R.O.C.
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan